CLINICAL TRIAL: NCT00358696
Title: TEN Switch - An Observational Phase IV Study to Evaluate the Safety and Efficacy of Substituting Tenofovir for Didanosine in Virologically Controlled HIV-infected Patients Co-infected With Hepatitis C Virus.
Brief Title: Antiretroviral Switch From Didanosine to Tenofovir in HIV/HCV Co-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Health Canada (Other Government)
Responsible Party: Dr. Brian Conway, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05-0218
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2009-10-20 (Estimated); Status verified 2009-10

CONDITIONS: HIV; HIV Infections
Keywords: tenofovir; didanosine; hiv; hepatitis c virus infection; treatment
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Hepatitis C | interventions — Tenofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: tenofovir — See Detailed Description.

SUMMARY:
The primary purpose of this study is to evaluate the impact of changing didanosine in an effective anti-HIV regimen to tenofovir on virologic suppression. We hypothesize that, in patients with maximal virologic suppression on a double class regimen (including two NRTIs and an NNRTI or a PI, boosted with RTV or not), a single drug substitution of didanosine for tenofovir will represent a viable strategy without any negative impact on the virologic efficacy of the regimen.

DETAILED DESCRIPTION:
Primary objective - to determine the impact of changing part of an effective HAART regimen to tenofovir on maintenance of virologic suppression in HCV co-infected patients.

Secondary objective - to assess the safety and tolerability over 12 weeks in patients switched to tenofovir.

Research Method - This will be a single arm observational study to include 30 subjects. Patients requiring HCV treatment will be assessed and patients receiving didanosine will be clinically evaluated to determine an appropriate NRTI drug switch. Patients who are to switch the didanosine component of their regimen to tenofovir will be eligible to participate in the study and will be followed for a period of observation of up to 4 weeks. All patients will be receiving tenofovir as one capsule, once daily. The primary endpoint will be maintenance of virologic suppression between the Baseline visit and week 12 in the overall study group. Measures of adherence to HAART, safety, tolerability and CD4 cell counts will also be obtained at each study visit, and will constitute secondary study endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. Be age 19 or older;
2. Have a confirmed diagnosis of HIV infection;
3. Have a confirmed positive HCV RNA PCR;
4. Have two consecutive HIV RNA levels <50 copies/mL with the most recent within the past 3 months;
5. Must not exhibit evidence of an acute illness, including an acute opportunistic infection;
6. Must not have any evidence of grade 3-4 laboratory abnormalities;
7. Must be able and willing to provide informed consent.

Exclusion Criteria:

1. Be receiving investigational drug within 30 days prior to beginning this study;
2. If female, be pregnant or breast-feeding;
3. In the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for participation for any reason.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-07; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Virologic Suppression

SECONDARY OUTCOMES:
HAART adherence, safety, CD4 cell count

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Brian Conway, MD, Principal Investigator — University of British Columbia
Locations (1):
- Pender Community Health Centre, Vancouver, British Columbia, Canada